CLINICAL TRIAL: NCT03960411
Title: Effect of Doxycycline on Cardiac Remodelling in Patients With ST-Elevation Myocardial Infarction (STEMI)
Brief Title: Effect of Doxycycline on Cardiac Remodelling in STEMI Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Felix Chikita Fredy, MD (Other)
Collaborators: National Cardiovascular Center Harapan Kita Hospital Indonesia (Other)
Responsible Party: Sponsor-Investigator, Felix Chikita Fredy, MD, cardiology resident, Indonesia University
Organization: Indonesia University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01
Record Dates: First submitted 2019-05-16; First posted 2019-05-23 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: ST Elevation Myocardial Infarction; Anterior Wall Myocardial Infarction; Heart Failure; Remodeling, Ventricular
Keywords: Doxycycline; Cardiac Remodelling; STEMI
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Anterior Wall Myocardial Infarction; Heart Failure; Ventricular Remodeling | interventions — Doxycycline

STUDY DESIGN:
Intervention Model Description: One arm receives standard care after primary PCI, the other receives doxycycline b.i.d for 7 days as an adjunct to standard care
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The only party who is not masked is the pharmacist
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Doxycycline (Experimental): Doxycycline 100 mg capsule by mouth every 12 hours for 7 days, administered early after primary PCI
  Interventions: Drug: Doxycycline 100Mg Capsule
- Placebo (Placebo Comparator): Placebo capsule by mouth every 12 hours for 7 days, administered early after primary PCI
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Doxycycline 100Mg Capsule — Doxycycline capsule
  Other Names: Doryx; Doxyhexal; Doxylin
  Arms: Doxycycline
Drug: Placebo oral capsule — Capsule manufactured to mimic doxycycline 100 mg capsule
  Other Names: Placebo (for Doxycycline)
  Arms: Placebo

SUMMARY:
Subsequent to the loss of myocardium post-myocardial infarction (MI), the affected ventricle undergoes some dynamic structural and functional changes known as remodeling. Cardiac remodeling progresses into heart failure (HF). In this revolutionized percutaneous coronary intervention (PCI) era, the incidence of post-MI HF due to cardiac remodeling remains high. Current standard therapeutic interventions, for HF, aimed solely at correcting a low cardiac output do not necessarily impede HF progression. Recently, doxycycline was found to have an additional biological effect aside from their antimicrobial actions. From several experimental studies and clinical trials, doxycycline showed MMP inhibition activities that can prevent ventricular remodeling. This study aims to evaluate the role of doxycycline in cardiac remodeling prevention post-MI. Our hypothesis is that a better heart function will be observed in STEMI patients who receive a short period of doxycycline administration post-PCI.

ELIGIBILITY:
Inclusion Criteria:

* Onset of STEMI <12 hours
* Anterior wall STEMI or Killip grade II-III or LVEF <50%
* Undergoing primary PCI

Exclusion Criteria:

* Signs of infection (clinical judgement plus leukocyte count >15,000)
* STEMI mechanical complication
* Moderate-severe valvular disease
* Allergic to doxycycline
* Refuse to join the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-05-25 (Actual); Primary Completion 2019-08 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
high sensitivity-Troponin T | 12 hours
  hs-Troponin T in ng/L
high sensitivity-CRP | 24 hours
  hs-CRP in mg/L
NT-pro BNP | 5 days
  NT-pro BNP in pg/ml
netrophils | 24 hours
  absolute amount per micro liters
ST2 | 24 hours
  ST2 in ng/ml

SECONDARY OUTCOMES:
Mortality rate | 4 months
  The number of deceased participants
Heart failure incidence | 4 months
  Evaluating the occurrence of heart failure signs and/or symptoms
Re-hospitalization rate | 4 months
  The number of patients re-admitted due to heart failure signs and/or symptoms
Left ventricle function and dimension | 4 months
  Assessed through echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Bambang Widyantoro, PhD, Principal Investigator — Indonesia University
Locations (1):
- National Cardiovascular Center Harapan Kita Hospital, Jakarta, Indonesia

REFERENCES:
- [Background] Cerisano G, Buonamici P, Valenti R, Sciagra R, Raspanti S, Santini A, Carrabba N, Dovellini EV, Romito R, Pupi A, Colonna P, Antoniucci D. Early short-term doxycycline therapy in patients with acute myocardial infarction and left ventricular dysfunction to prevent the ominous progression to adverse remodelling: the TIPTOP trial. Eur Heart J. 2014 Jan;35(3):184-91. doi: 10.1093/eurheartj/eht420. Epub 2013 Oct 8. PMID 24104875